CLINICAL TRIAL: NCT04025320
Title: The Effect of Intraneural Facilitation Therapy on Diabetic Patients With Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Lee Berk, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5190128
Record Dates: First submitted 2019-06-11; First posted 2019-07-18 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Intraneural facilitation treatment for 50-60 minutes. 50 minutes if ultrasound received.
  9 total treatment visits, 3 visits per week
  • One 50-60 minute visit on Monday, Wednesday and Friday, for 3 weeks.
  Interventions: Other: Intraneural Facilitation
- Group 2 (Sham Comparator): SHAM treatment for 50-60 minutes. 50 minutes if ultrasound received. 9 total treatment visits, 3 visits per week
  • One 50-60 minute visit on Monday, Wednesday and Friday, for 3 weeks.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Intraneural Facilitation — Intraneural Facilitation utilizes three manual holds. Firstly, the contralateral joint is placed in a maximal loose-pack position to pressurize the nervous system and bias circulation from the artery into the epineurium. Now that we have increased this pressure we begin the secondary hold to bias the increased epineurial blood into the transperineurial vessels that bridge the epiperineum and the endoneurial capillaries of the site being treated. Now that the pressure has increased into the open endoneurial capillaries, the goal is to open up ischemic endoneurial capillaries and this is hypothesized to open by providing the third hold. The third hold is known as the sub hold and encourages blood flow through ischemic endoneurial capillaries that have increased resistance/pressure through the application of bernoulli's principle. This treatment will take 50-60 minutes.
  Arms: Group 1
Other: Sham — A physical therapist will perform the SHAM light therapy at the same site as the INF therapy location, at the Neuropathic Treatment Center. The SHAM light therapy will last 50-60 minutes and consists of using an anodyne unit for application of near-infrared light therapy. The unit will not be switched on, but the pads will be placed on the subject and the subject will be blinded to the unit being on. The anodyne therapy pads will be placed in the following locations on the affected lower limb: two on the plantar aspect of the foot in a T formation and one pad on the medial and lateral side of the calf. A double folded towel will be wrapped around the subject's foot at the electrode sites to blind the subject's from the light not emitting from the electrodes, due to the anodyne unit being off.
  Arms: Group 2

SUMMARY:
The purpose of this graduate student research study is to explore the effects of a new treatment known as Intraneural facilitation (INF) on Diabetes Mellitus Type 2 (DMT2) subjects who have moderate - severe below ankle neuropathy symptoms. Since INF has shown success in the clinic and significant improvements have been found in a recent pilot study, this study aims to further explore these effects on DMT2 subjects suffering from DPN. The investigators would like to investigate if INF improves blood flow in the foot, if it decreases the pain and improves the sensation, and if it improves the overall quality of life.

DETAILED DESCRIPTION:
The demographic data (age, height, gender, and weight) will be collected from each subject. All subjects will go through the following protocol: First, subjects will complete pre-testing measurements consisting of 5 tests; Pain Quality Assessment Scale, Semmes-Weinstein Monofilaments, NeuroCom SMART Balance Master, Quality of Life- Diabetic Neuropathy Scale (QOL- DN), and Zeno Walkway. Patients will then be randomized into two groups and blinded by the treatment. Patients who draw "Group 1" will be given the INF treatment and patients who draw "Group 2" will be given the SHAM treatment. Patients will then be completing 3 weeks of INF treatment, or SHAM treatment for 3 visits per 3 week, totaling 9 treatment visits. Post treatment, patients will then return for the same 5 measurements completed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Type 2 and Diabetic Peripheral Neuropathy with no other known underlying disease
* Below ankle Diabetic Peripheral Neuropathy symptoms (numbness, tingling, burning, sharp pain, increased sensitivity, etc.)
* ≥10 on Quality of Life- Diabetic Neuropathy Scale (QOL- DN)
* Between age 50-75 years

Exclusion Criteria:

* Patients with a medical condition that suggested possible decline in function over the next 6 months such as; a current regimen of chemotherapy, radiation therapy, or dialysis
* Any lower extremity amputations or wounds
* Documented active alcohol and/or drug misuse
* Known health conditions: end stage renal failure, uncontrolled hypertension, severe dyslipidemia, chronic liver disease, autoimmune disease, advanced chronic obstructive pulmonary disease and active inflammations
* DM patients with inflammatory neuropathies including chronic inflammatory demyelinating polyneuropathy (CIDP), proximal diabetes neuropathy, and autonomic neuropathies
* Patients with other types of neuropathies not associated with Diabetes Mellitus such as B12 deficiency, hypothyroidism, and uremia
* Other severe chronic medical condition requiring active treatment
* Morbidly Obese patients
* Pregnancy (self reported)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Pain Quality Assessment Scale | change between baseline and 5 weeks
  It is a self-report tool derived from Neuropathic Pain Scale to evaluate the quality of neuropathic pain. After reading the introduction of the questionnaire, subjects will then measure their pain on a numeric scale 0= "no pain" or "no painful sensation" to 10 = "worst imaginable pain sensation" . A zero score represents the best outcome and a 10 is the worst outcome. This questionnaire takes approximately 10 minutes.

SECONDARY OUTCOMES:
Limits of Stability | change between baseline and 5 weeks
  The LOS test will assess the subjects weight-shifting ability and voluntary limits of stability to eight directional targets set at 100% of theoretical limits of stability for an eight second hold. The LOS test measures five parameters: reaction time, movement velocity, end point excursion, maximum excursion, and directional control. We will take the composite scores of reaction time, movement velocity, end point excursion, maximum excursion, and directional control from the 8 directions. This test should take 10 minutes.
Zeno Walkway | change between baseline and 5 weeks
  The Zeno Walkway is used to observe the spatiotemporal characteristics of gait in the subjects: velocity and stride length. Participants will be wearing their own shoes and will be instructed prior to arrival to wear comfortable shoes without heels. The subjects will be asked to walk back and forth the walkway 4 times. This test will take 5 minutes.
Sensory organization test (SOT) | change between baseline and 5 weeks
  The SOT will assess the subject's use of visual, somatosensory, and vestibular systems for maintaining upright posture. The standardized test instructions, per NeuroCom protocol, were either "stand quietly with your eyes open" or "stand quietly with your eyes closed" depending on the condition being tested. This test is completed under six different sensory conditions lasting 20 seconds each.
  * Step 1 the patient is required to stand still with eyes open (all sensory information available)
  * Step 2 the patient is required to stand still with their eyes closed
  * Step 3 the surrounding moves as the patient moves
  * Step 4 the force plate moves as the patient moves
  * Step 5 the patient closes their eyes and the force plate moves as the patient moves
  * Step 6 the surrounding and force plate move as the patient moves This test should take 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Berk, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

REFERENCES:
- [Derived] Sahba K, Berk L, Bussell M, Lohman E, Zamora F, Gharibvand L. Treating peripheral neuropathy in individuals with type 2 diabetes mellitus with intraneural facilitation: a single blind randomized control trial. J Int Med Res. 2022 Aug;50(8):3000605221109390. doi: 10.1177/03000605221109390. PMID 35922961